CLINICAL TRIAL: NCT00476957
Title: PROTECT Trial: Patient Related OuTcomes With Endeavor Versus Cypher Stenting Trial
Brief Title: Randomized Study Comparing Endeavor With Cypher Stents (PROTECT)
Acronym: PROTECT
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Medtronic Vascular (Industry)
Collaborators: Medtronic Cardiac Rhythm and Heart Failure (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Health Services Research
Other Study IDs: Version 1.0 - 12 April 2007
Record Dates: First submitted 2007-05-21; First posted 2007-05-22 (Estimated); Results first posted 2014-03-17 (Estimated); Last update posted 2014-11-10 (Estimated); Status verified 2014-11

CONDITIONS: Ischemic Heart Disease
Keywords: Drug Eluting Stents; Interventional Cardiology
MeSH Terms: conditions — Myocardial Ischemia | interventions — Stents

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- 1 (Active Comparator): Medtronic Endeavor® Zotarolimus Eluting Coronary Stent System
  Interventions: Device: Stent
- 2 (Active Comparator): Cordis Cypher® Sirolimus-eluting Coronary Stent
  Interventions: Device: Stent

INTERVENTIONS:
Device: Stent — Stent implantation
  Other Names: Medtronic Endeavor® Zotarolimus Eluting Coronary Stent System
  Arms: 1
Device: Stent — Stent implantation
  Other Names: Cordis Cypher® Sirolimus-eluting Coronary Stent
  Arms: 2

SUMMARY:
The PROTECT TRIAL is a randomized stent trial with 8800 patients in approximately 200 hospitals, which is designed to evaluate whether the Endeavor stent PROTECTS against late stent thrombosis resulting in less deaths and myocardial infarctions.

Study Stents:

Medtronic Endeavor® Zotarolimus Eluting Coronary Stent System or next generation model Cordis Cypher® Sirolimus-eluting Coronary Stent, Cordis Cypher Select® Sirolimus-eluting Coronary Stent or next generation model

Primary Objective: To compare overall stent thrombosis rate of the Endeavor® Zotarolimus Eluting Coronary Stent System versus the Cypher® Sirolimus-eluting Coronary Stent in a patient population requiring stent implantation

Secondary Objective: To compare the composite endpoint of total death or cardiac death combined with the number of patients with all non-fatal myocardial infarctions as well as the number of patients with large non-fatal myocardial infarctions for Endeavor® Zotarolimus Eluting Coronary Stent System versus the Cypher® Sirolimus-eluting Coronary Stent in a patient population requiring stent implantation.

To assess the safety and efficacy in patient subgroups with specific demographics, clinical indications and/or vessel- or lesion characteristics.

ELIGIBILITY:
Inclusion Criteria:

1. Patient is > 18 years of age (or minimum age as required by local regulations).
2. The patient has consented to participate and has authorized the collection and release of his medical information by signing the "Patient Informed Consent Form".
3. All lesions requiring interventions (target lesions - one to a maximum of four) in one or more native coronary arteries are amendable for implantation of one or more Endeavor® Zotarolimus Eluting Coronary Stent System or Cypher® Sirolimus-eluting Coronary Stent*.
4. Patient indication, lesion length and vessel diameter of the target lesion(s) are according to the 'Indications for Use' as mentioned in the 'Instructions for Use' that comes with every Endeavor® Zotarolimus Eluting Coronary Stent System and Cypher® Sirolimus-eluting Coronary Stent. Patients should qualify for both systems before randomization*.
5. The patient is willing and able to cooperate with study procedures and required follow up visits.

Exclusion Criteria:

1. Women with known pregnancy or who are lactating.
2. Planned elective surgery necessitating discontinuation of clopidogrel within the regular planned period of clopidogrel administration.
3. Patients expected not to be compliant with the anti-platelet and/or anticoagulation therapy regimen.
4. Previous brachy-therapy.
5. Previous implantation of a drug eluting stent.
6. Previous implantation of a bare metal stent in the preceding year.
7. Simultaneous or planned intervention other non cardiac vessels including but not limited to renal artery or carotid artery.
8. Current medical condition with a life expectancy of less than 3 years.
9. Manifest acute severe heart failure (Killip class III-IV).
10. The patient is currently, and during the first 3 years of the PROTECT trial, participating in another investigational device or drug study that clinically interferes with the PROTECT-study endpoints; or requires coronary angiography or other coronary artery imaging procedures. The patient may only be enrolled in the PROTECT-study once.
11. Patients with medical conditions that preclude the follow-up as defined in the protocol or that otherwise limits participation in this study.
12. Patients on warfarin or similar anti-coagulant therapy.
13. Patients with hypersensitivity or allergies to one of the drugs or components indicated in the Instructions for Use of either stents.
14. Patients who are judged to have a lesion that prevents complete inflation of an angioplasty balloon.
15. Patients in whom anti-platelet and/or anticoagulation therapy is contraindicated.
16. Transplant patients.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 8709 (Actual)
Dates: Start 2007-06; Primary Completion 2012-05 (Actual); Study Completion 2014-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Edoardo Camenzind, MD, Principal Investigator — University of Geneva, Switzerland; Laura Mauri, MD, Principal Investigator — Brigham and Women's Hospital, US; William O'Neill, MD, Principal Investigator — University of Miami Miller School of Medicine, US; Prof. Patrick W. Serruys, MD, PhD, Principal Investigator — Erasmus Medical Center; Prof. Philippe Gabriel Steg, MD, PhD, Principal Investigator — Département de Cardiologie, Hôpital Bichat-Claude Bernard, Assistance Publique - Hôpitaux de Paris, France; William Wijns, MD, PhD, Principal Investigator — O.L.V. Hospital, Aalst, Belgium
Locations (1):
- 196 enrolling sites Worldwide, Maastricht, Netherlands

REFERENCES:
- [Background] Camenzind E, Wijns W, Mauri L, Boersma E, Parikh K, Kurowski V, Gao R, Bode C, Greenwood JP, Gershlick A, O'Neill W, Serruys PW, Jorissen B, Steg PG; PROTECT Steering Committee and Investigators. Rationale and design of the Patient Related OuTcomes with Endeavor versus Cypher stenting Trial (PROTECT): randomized controlled trial comparing the incidence of stent thrombosis and clinical events after sirolimus or zotarolimus drug-eluting stent implantation. Am Heart J. 2009 Dec;158(6):902-909.e5. doi: 10.1016/j.ahj.2009.10.002. PMID 19958855
- [Result] Camenzind E, Wijns W, Mauri L, Kurowski V, Parikh K, Gao R, Bode C, Greenwood JP, Boersma E, Vranckx P, McFadden E, Serruys PW, O'Neil WW, Jorissen B, Van Leeuwen F, Steg PG; PROTECT Steering Committee and Investigators. Stent thrombosis and major clinical events at 3 years after zotarolimus-eluting or sirolimus-eluting coronary stent implantation: a randomised, multicentre, open-label, controlled trial. Lancet. 2012 Oct 20;380(9851):1396-405. doi: 10.1016/S0140-6736(12)61336-1. Epub 2012 Aug 27. PMID 22951082
- [Derived] Roguin A, Camenzind E, Kerner A, Beyar R, Boersma E, Mauri L, Steg PG, Wijns W. Long-Term Outcomes of Stenting the Proximal Left Anterior Descending Artery in the PROTECT Trial. JACC Cardiovasc Interv. 2017 Mar 27;10(6):548-556. doi: 10.1016/j.jcin.2016.12.028. PMID 28335893
- [Derived] Secemsky EA, Matteau A, Yeh RW, Steg PG, Camenzind E, Wijns W, McFadden E, Mauri L; PROTECT Trial Investigators. Comparison of Short- and Long-Term Cardiac Mortality in Early Versus Late Stent Thrombosis (from Pooled PROTECT Trials). Am J Cardiol. 2015 Jun 15;115(12):1678-84. doi: 10.1016/j.amjcard.2015.03.010. Epub 2015 Mar 23. PMID 25910523
- [Derived] Wijns W, Steg PG, Mauri L, Kurowski V, Parikh K, Gao R, Bode C, Greenwood JP, Lipsic E, Alamgir F, Rademaker-Havinga T, Boersma E, Radke P, van Leeuwen F, Camenzind E; PROTECT Steering Committee and Investigators. Endeavour zotarolimus-eluting stent reduces stent thrombosis and improves clinical outcomes compared with cypher sirolimus-eluting stent: 4-year results of the PROTECT randomized trial. Eur Heart J. 2014 Oct 21;35(40):2812-20. doi: 10.1093/eurheartj/ehu318. Epub 2014 Aug 8. PMID 25106761
- [Derived] Camenzind E, Boersma E, Wijns W, Mauri L, Rademaker-Havinga T, Ordoubadi FF, Suttorp MJ, Al Kurdi M, Steg PG; PROTECT Steering Committee and Investigators. Modifying effect of dual antiplatelet therapy on incidence of stent thrombosis according to implanted drug-eluting stent type. Eur Heart J. 2014 Aug 1;35(29):1932-48. doi: 10.1093/eurheartj/ehu084. Epub 2014 Mar 13. PMID 24627416

RESULTS

PARTICIPANT FLOW:
Recruitment Details: 8709 patients were randomized from May 2007 until December 2008 in 196 participating hospitals in 36 countries across five continents.
Pre-assignment Details: 80 patients were excluded because there was no validly signed consent available during monitoring and 2 patients retracted their consent before the procedure, resulting in a total of 8709 patients randomised.
Groups:
- E-ZES: Medtronic Endeavor® Zotarolimus Eluting Coronary Stent System
  Stent : Stent implantation
- C-SES: Cordis Cypher® Sirolimus-eluting Coronary Stent
  Stent : Stent implantation
Period: Overall Study
Arm/Group | E-ZES | C-SES
Started | 4357 | 4352
Completed | 4181 | 4159
Not Completed | 176 | 193
Not completed — Lost to Follow-up | 176 | 193

BASELINE CHARACTERISTICS:
Population: Intention to treat analysis has been used.
Groups:
- Total: Total of all reporting groups
Arm/Group | E-ZES | C-SES | Total
Number analyzed (Participants) | 4357 | 4352 | 8709
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 2428 | 2468 | 4896
  >=65 years | 1929 | 1884 | 3813
Age, Continuous [Mean (Standard Deviation); unit: years] | 62.3 (10.6) | 62.1 (10.7) | 62.2 (10.6)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1017 | 1044 | 2061
  Male | 3340 | 3308 | 6648
Region of Enrollment [Number; unit: participants]
  Europe | 3180 | 3179 | 6359
  South Asia | 623 | 622 | 1245
  North America | 115 | 115 | 230
  South America | 25 | 25 | 50
  Australia | 207 | 207 | 414
  New Zealand | 43 | 42 | 85
  Middle East | 164 | 162 | 326

OUTCOME MEASURES:

1. Primary Outcome: To Compare Overall Definite or Probable Stent Thrombosis Rate of the Endeavor® Zotarolimus Eluting Coronary Stent System Versus the Cypher® Sirolimus-eluting Coronary Stent in a Patient Population Requiring Stent Implantation
Description: Definite or probable stent thrombosis rate.
Time Frame: 3 years
Measure: Number; unit: participants
Arm/Group | E-ZES | C-SES
Number analyzed (Participants) | 4357 | 4352
participants | 61 | 75

2. Secondary Outcome: Composites of (Cardiac) Death and (Large) Non-fatal Myocardial Infarctions
Description: Total death and large non-fatal myocardial infarctions Total death and non-fatal myocardial infarctions Cardiac death and large non-fatal MI Cardiac death and non-fatal myocardial infarctions
Time Frame: 3 years
Measure: Number; unit: participants
Arm/Group | E-ZES | C-SES
Number analyzed (Participants) | 4357 | 4352
participants
  Total death and large non-fatal myocardial infarct | 225 | 255
  Total death and non-fatal myocardial infarctions | 331 | 360
  Cardiac death and large non-fatal MI | 157 | 174
  Cardiac death and non-fatal MI | 265 | 282
  Target lesion revascularization | 249 | 156
  Stroke | 77 | 72
  Bleeding events | 201 | 184

ADVERSE EVENTS:
Arm/Group | E-ZES | C-SES
Serious Adverse Events (participants affected / at risk) | 579/4357 | 507/4352
Other Adverse Events (participants affected / at risk) | 201/4357 | 184/4352
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | E-ZES (N=4357) | C-SES (N=4352)
MACCE (major adverse cardiac and cerebrovascular event (Cardiac disorders) | 579 (579) | 507 (507)
OTHER ADVERSE EVENTS (reported when occurring in more than 4.6% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | E-ZES (N=4357) | C-SES (N=4352)
Bleeding (Blood and lymphatic system disorders) | 201 (201) | 184 (184)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
For any publication or presentation of the Protected Materials or any portion thereof, a manuscript of the paper, abstract or other materials will be provided by Consultant to Sponsor for its approval at least sixty (60) days for manuscripts and thirty (30) days for presentations prior to outside submission. Medtronic shall have the right to request reasonable modifications of any manuscript or other materials to be published or presented.